CLINICAL TRIAL: NCT04896619
Title: Cholesterol Effects of Kori-tofu Proteins
Acronym: CHOKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: Asahimatsu Foods (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NL75320.081.20
Record Dates: First submitted 2021-05-10; First posted 2021-05-21 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Lipid Metabolism Disorders
Keywords: Kori tofu; Cholesterol
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily dose of Kori-tofu mixed in 3 slices of bread (Experimental): Kori tofu as part of bread
  Interventions: Other: Kori tofu bread
- Daily dose of whey protein, soy oil and maltodextrin mixed in 3 slices of bread (Active Comparator): Whey protein, soy oil and maltodextrin as part of bread
  Interventions: Other: Whey protein bread

INTERVENTIONS:
Other: Kori tofu bread — 34.5 grams of Kori-tofu, mixed in 3 slices of wheat bread.
  Arms: Daily dose of Kori-tofu mixed in 3 slices of bread
Other: Whey protein bread — Matched whey protein, soy oil and maltodextrin/cellulose, mixed in 3 slices of wheat bread
  Arms: Daily dose of whey protein, soy oil and maltodextrin mixed in 3 slices of bread

SUMMARY:
The study is a randomized, cross-over, double-blind, controlled trial in which participants with mildly elevated levels of cholesterol will receive two 4-week interventions (e.g. kori-tofu or control), with a wash-out period of 4 weeks in between. During the intervention periods, subjects will eat 3 slices of bread per day, representing a Kori-tofu dose of 34.5 grams or a matched reference. Fasting total and LDL cholesterol will be determined at the start and end of each of the two intervention periods.

DETAILED DESCRIPTION:
There are several types of tofu, an example of a specific type of tofu is called Kori-tofu. Kori-tofu literally means frozen tofu. The production process of Kori-tofu leads to the formation of a higher high molecular weight fraction (HMF) content of the soy proteins. Several studies describe the effects of Kofi-tofu on health. In this study the aim is to investigate the effect of repetitive consumption of Kori-tofu on blood cholesterol levels and other lipid metabolism related measures, in research subjects with mildly elevated levels of cholesterol.

The primary objective is to assess the effect of repetitive consumption of Kori-tofu on blood total and LDL cholesterol levels. The secondary objective is to assess the effect of repetitive consumption of Kori-tofu on other markers of lipid metabolism, glucose metabolism and blood pressure.

The study is a randomized, cross-over, double-blind, controlled trial in which participants will receive two 4-week interventions (e.g. kori-tofu or control), with a wash-out period of 4 weeks in between. During the intervention periods, subjects will eat 3 slices of bread per day, representing a Kori-tofu dose of 34.5 grams or a matched reference (whey protein, soy oil and maltodextrin/cellulose). Research subjects will visit our research unit before and after each intervention period for a test day. During these test days fasting blood samples will be collected and blood pressure measurements will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-70 years;
* BMI between 18.5-35 kg/m2;
* Total cholesterol levels >5 mmol/L or LDL >3 mmol/L

Exclusion Criteria:

* Use of medication/supplements/food items that may influence the study results, such as cholesterol lowering medication, Becel ProActiv (judged by our research physician);
* Total cholesterol levels >7 mmol/L;
* LDL cholesterol levels >5 mmol/L;
* Reported slimming, medically prescribed or other extreme diets;
* Reported weight loss or weight gain of >5 kg in the month prior to pre-study screening;
* Not willing to give up blood donation during the study;
* Current smokers;
* Alcohol intake ≥4 glasses of alcoholic beverages per day;
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported);
* Abuse of soft and/or hard drugs;
* Food allergies or intolerances for products that we use in the study;
* Participation in another clinical trial at the same time; NL75320.081.20 CHOKO Version number: 4, April 2021 15 of 34
* Being an employee of the Food, Health & Consumer Research group of Wageningen Food & Biobased Research.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Change in total cholesterol levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in LDL cholesterol levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions

SECONDARY OUTCOMES:
Change in HDL cholesterol levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in triglycerides levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in leptin levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in adiponectin levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in plasma insulin levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in HbA1c levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in fructosamine levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in glucose levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in systolic blood pressure levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions
Change in diastolic blood plessure levels | 0 weeks, 4 weeks, 8 weeks and 12 weeks
  under fasting conditions

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University & Research
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No